CLINICAL TRIAL: NCT01019005
Title: Pain Relief After Forefoot Surgery: Tibial Perineural Catheter vs. Wound Catheter Infusion
Brief Title: Pain Relief After Forefoot Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Nottingham University Hospitals NHS Trust, Queens' Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QMC-1975-HJ; QMC-1975-NB (Other: QMC)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Orthopedic Surgery
Keywords: post-operative analgesia; opioid; catheter; tibial nerve block
MeSH Terms: interventions — Catheters

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tibial (Experimental)
  Interventions: Device: Catheter
- Wound (Experimental)
  Interventions: Device: Catheter
- Sham (No Intervention)
  Interventions: Device: Catheter

INTERVENTIONS:
Device: Catheter — Catheter inserted into either perineural tibial nerve or wound

SUMMARY:
The aim to test whether continues local anaesthetic infusion via tibial catheter or wound catheter will improve pain relief following forefoot surgery

In this sequential prospective randomised, controlled clinical trial,75 Patients undergoing forefoot surgery will be randomized into three groups (tibial, wound, control). All groups will receive ankle block ± general anesthetic (standard technique). The tibial group will have a tibial catheter inserted through which local anaesthetic will be infused. The wound group will have a catheter inserted directly into the wound immediately after surgery. The control group will have a sham catheter (covered by a bandage across foot) attached to a pump which will not infuse. Patient maximum pain scores (primary outcome measure), nausea/ vomiting, analgesia use, satisfaction and sleep disturbance will be recorded postoperatively. All groups will be then followed by telephone calls 48 hours. Patients will be instructed to come to the clinic on the 4th postoperative day where the catheter will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older (ASA I & II)
* Able to give written consent
* Patients having elective forefoot surgery with a planned ankle block.
* Expected postoperative pain to be at least moderate in severity the day following surgery

Exclusion Criteria:

* Refusal
* Inability to communicate
* History of alcohol or opioid abuse (also chronic opioid user)
* Mental or medical conditions which may affect quantifying pain scores (VAS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 2,8,12,24,48 hr

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom